CLINICAL TRIAL: NCT07264114
Title: The Effect of Aquatic High-Intensity Interval Training on Balance, Physical Function, and Sarcopenia in Patients With Parkinson's Disease: A Randomized Controlled Trial Protocol
Brief Title: Aquatic High-Intensity Interval Training for Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PA25PKD-2-01
Record Dates: First submitted 2025-11-18; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Aquatic Exercise; High-Intensity Interval Training; Balance; Sarcopenia; Quality of Life; Sleep Quality
MeSH Terms: conditions — Parkinson Disease; Sarcopenia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocate to intervention group or control group and will be examined in the same way.
Masking Description: None (Open Label) for participants and care providers; Single (Outcomes Assessor) for functional tests; Blinded data analysis."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic HIIT group (Experimental): The participants in the experimental group will undertake supervised aquatic high-intensity interval exercise 3×/week for 8 weeks (Tabata method). Each session consists of a 10-min warm-up, Tabata sets (20s maximal-effort aquatic exercises-e.g., water running, jumping jacks, resistance with foam dumbbells/paddles-followed by 10s rest, 8 cycles/set; total set=4 min), and a 5-min cool-down.
  Intensity monitored using Borg RPE scale (6-20), target 15-17 ("hard" to "very hard") during work phases to ensure HIIT delivery. RPE recorded at end of each set with real-time feedback (e.g., "push harder" if <15). Validated in PD trials; RPE 15-17 ≈80-90% max HR in water (HR optional).
  Pool depth waist-to-chest (≈1.2-1.4 m), temp 32-34 °C. Delivered in indoor therapeutic pool of Pardis Institute by certified specialists. Standard medical care continues. Adherence via attendance logs; >20% missed = non-adherent.
  Interventions: Behavioral: Aquatic HIIT with adherence/support package
- Control group (No Intervention): Patients allocated to the control group will receive their usual clinical management for Parkinson's disease, including pharmacological therapy as prescribed by their neurologist, and will not participate in any structured exercise program during the 8-week study period. Low-intensity daily activities and usual physical routines are permitted. Control participants will be advised to maintain their standard treatment regimen and customary activity patterns during the trial.

INTERVENTIONS:
Behavioral: Aquatic HIIT with adherence/support package — The participants in the behavioral component will receive the same supervised aquatic HIIT program described above plus structured behavioral/support measures to maximize adherence and safety. These include: an initial individual education session explaining benefits/risks and protocol; supervised real-time feedback during each session from exercise specialists; flexible scheduling options to accommodate participants; weekly review of attendance and brief motivational follow-up (phone call or in-person) for participants with missed sessions; individualized adjustments to intensity/duration based on participant feedback and safety; and documentation of reasons for non-attendance. All behavioral/support activities are delivered by trained research staff and exercise physiologists and are recorded in session logs. (These measures are drawn from the protocol's adherence and retention strategies.)
  Arms: Aquatic HIIT group

SUMMARY:
This randomized, single-center, parallel-group superiority trial will evaluate the effect of an 8-week aquatic High-Intensity Interval Training (HIIT) program on balance, physical function, and sarcopenia-related outcomes in individuals with Parkinson's disease (PD). The intervention aims to deliver Tabata-style aquatic HIIT (3 sessions/week) in a therapeutic pool to determine adherence and preliminary efficacy compared with standard care (no structured exercise program).

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by motor and non-motor symptoms that impair quality of life. Pharmacological treatments alleviate motor symptoms but leave residual motor and non-motor complications and carry long-term adverse effects. Non-pharmacological therapies-particularly exercise-improve motor and non-motor outcomes via mechanisms such as enhanced dopamine release, corticostriatal plasticity, and increased BDNF after vigorous exercise. HIIT (including Tabata protocols) has emerging evidence for benefit in PD but land-based HIIT can be limited by balance deficits and fall risk. Aquatic HIIT may provide a safer environment (buoyancy, reduced joint load, natural resistance) and improve adherence.

This single-center trial will recruit 56 participants (aged 55-75) with PD (Hoehn & Yahr stages 2-3) and balance difficulty to be randomized 1:1 to aquatic HIIT (n=28) or control (standard care; n=28). The intervention comprises 8 weeks of supervised Tabata-format aquatic sessions (20s high intensity/10s rest ×8 cycles per set; warm-up and cool-down included) three times weekly. Primary endpoints include changes in Berg Balance Scale (BBS), Short Physical Performance Battery (SPPB), skeletal muscle mass by BIA, and handgrip strength from baseline to Week 8 (primary endpoint), with safety follow-up to Week 12. Secondary endpoints include PDQ-39, PSQI, adherence, and adverse events monitored with CTCAE criteria.

ELIGIBILITY:
Inclusion Criteria:

* PD stages 2-3 based on Hoehn and Yahr classification system
* Balance difficulty (BBS score <45)
* Reduced motor function
* Sarcopenia (per EWGSOP2 criteria)
* Age ≥ 55
* Permission from their doctors to participate
* Absence of a history of myocardial infarction within the past 3 months
* Capacity to provide informed consent to participate in the study

Exclusion Criteria:

* Cardiac instability (angina, decompensated congestive heart failure, severe arteriovenous stenosis, uncontrolled arrhythmias, etc.)
* Active infection or acute medical illness
* Hemodynamic instability
* Labile glycemic control
* Inability to exercise (e.g. lower extremity amputation with no prosthesis)
* Severe musculoskeletal pain at rest or with minimal activity
* Inability to sit, stand or walk unassisted (walking device such as cane or walker allowed)
* Shortness of breath at rest or with activities of daily living

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Rate of changes in Balance Ability | Pre-intervention and Week 8
  Evaluating the effect of aquatic HIIT on balance using the Berg Balance Scale (BBS), a 14-item performance-based tool assessing static and dynamic balance through functional tasks like sitting to standing, reaching forward, and turning 360 degrees. Items are scored on a 5-point ordinal scale (0-4) based on ability and time to complete, with a total score ranging from 0 (worst) to 56 (best); scores of 0-20 indicate wheelchair-bound, 21-40 indicate walking with assistance, and 41-56 indicate independent. In PD, scores <45 suggest high fall risk, and the BBS has excellent intra-rater reliability (ICC=0.98), inter-rater reliability (ICC=0.97), and criterion validity, correlating with other PD-specific measures like UPDRS.
Rate of changes in Physical Function | Pre-intervention and Week 8
  Evaluating the effect of aquatic HIIT on physical function using the Short Physical Performance Battery (SPPB), a composite test including three subcomponents: balance (holding side-by-side, semi-tandem, and tandem stands for up to 10 seconds each, scored 0-4), gait speed (timed 4-meter walk at usual pace, scored 0-4 based on time quartiles), and chair stand (time to complete five rises from a chair without arms, scored 0-4). Total score ranges from 0 (worst) to 12 (best), with scores <10 indicating high risk for mobility limitations and falls in older adults, including PD patients. The SPPB demonstrates high test-retest reliability (ICC=0.92), intra-rater reliability, and validity in predicting functional decline and executive function associations in PD.
Rate of changes in Muscle Mass (Sarcopenia) | Pre-intervention and Week 8
  Evaluating the effect of aquatic HIIT on sarcopenia-related muscle mass using Bioelectrical Impedance Analysis (BIA), a non-invasive technique that estimates body composition by measuring resistance and reactance to a low-level electrical current, calculating skeletal muscle mass (ASM) and phase angle (PhA). ASM is indexed to height squared (ASM/height² in kg/m²), with sarcopenia diagnosed per EWGSOP2 criteria (<7.0 kg/m² for men, <5.5 kg/m² for women); PhA cut-offs for sarcopenia are ≤4.05° (92.9% sensitivity, 53.8% specificity) for men and ≤3.75° (78.9% sensitivity, 51.1% specificity) for women. In PD, BIA is reliable for detecting sarcopenia (prevalence 40-55%) with high correlation to dual-energy X-ray absorptiometry (DXA) as gold standard (r=0.85-0.90 for ASM), predictive validity (adjOR=0.147 for PhA), and good test-retest reliability (ICC=0.88-0.95), though wide diagnostic variations exist across criteria.
Rate of changes in Muscle Strength | Pre-intervention and Week 8
  Evaluating the effect of aquatic HIIT on muscle strength using a Handgrip Dynamometer, a handheld device that quantifies isometric grip force in kilograms or pounds during maximal voluntary contraction (typically 3 trials per hand, with the highest or average value used). Measurements are taken in a standardized seated position with the elbow flexed at 90 degrees; normative values decline with age, and low grip strength (<27 kg men, <16 kg women) is a sarcopenia criterion in PD. The dynamometer shows fair to excellent test-retest reliability (ICC=0.95-0.98) and intra-rater reliability in PD, with good validity for overall strength assessment.

SECONDARY OUTCOMES:
Change in Quality of Life | Pre-intervention and Week 8
  Evaluating improvements in quality of life using the Parkinson's Disease Questionnaire-39 (PDQ-39), a disease-specific 39-item self-report instrument covering eight domains (mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, bodily discomfort). Items are rated on a 5-point Likert scale (0=never to 4=always), with domain scores transformed to 0-100 (higher indicating worse quality of life) and a summary index as the mean. The PDQ-39 has strong convergent validity (correlates with EQ-5D), discriminant validity, internal consistency (Cronbach's alpha=0.51-0.96), and test-retest reliability (0.56-0.90 per domain) in PD.
Change in Sleep Quality | Pre-intervention and Week 8
  Evaluating changes in sleep quality using the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-report questionnaire (plus 5 roommate-rated items) assessing seven components (subjective quality, latency, duration, efficiency, disturbances, medication use, daytime dysfunction) over the past month. Global score sums to 0-21 (higher=worse sleep), with >5 indicating poor quality (prevalence ~85% in PD). The PSQI has good internal consistency (Cronbach's alpha=0.83), test-retest reliability (0.85), and validity in PD, correlating with PSG and other scales like PDSS.
Adherence Rate | Week 0 to Week 8 (intervention period)
  Determining adherence to the intervention using attendance logs, which record session participation as a percentage (number of attended sessions / total planned sessions; Adherence defined as attending ≥80% of sessions (≤20% missed)."). Logs also note reasons for non-attendance, providing qualitative insights. This method is reliable for monitoring exercise adherence in PD trials, with group rates often >80% in supervised programs, though individual accuracy requires caution.
Adverse Events | Week 0 to Week 12 (including 4-week follow-up)
  Monitoring and reporting adverse events using the Common Terminology Criteria for Adverse Events (CTCAE v5.0 or later), a standardized system categorizing events by organ system and severity grades (1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death-related). Events are defined as any unfavorable sign, symptom, or disease temporally associated with the intervention; serious events (grades 3-5) prompt reporting to DSMB. CTCAE ensures consistent AE reporting in clinical trials, with updates like v6.0 in 2025.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Tabibi, Dr, Study Director — Pardis Specialized Wellness Institute

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the published article, after deidentification are to be shared
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available starting 6 months after publication of primary results (anticipated March 2026). No end date.
Access Criteria: Not applicable. It will be accessible for public.

REFERENCES:
- [Background] Harpham C, Gunn H, Marsden J, Bescos Garcia R, Connolly L. Home-based high-intensity interval training for people with Parkinson's: Protocol for the HIIT-Home4Parkinson's randomized, controlled feasibility study. Health Sci Rep. 2024 Jan 7;7(1):e1800. doi: 10.1002/hsr2.1800. eCollection 2024 Jan. PMID 38192731
- [Background] Kathia MM, Duplea SG, Bommarito JC, Hinks A, Leake E, Shannon J, Pitman J, Khangura PK, Coates AM, Slysz JT, Katerberg C, McCarthy DG, Beedie T, Malcolm R, Witton LA, Connolly BS, Burr JF, Vallis LA, Power GA, Millar PJ. High-intensity interval versus moderate-intensity continuous cycling training in Parkinson's disease: a randomized trial. J Appl Physiol (1985). 2024 Sep 1;137(3):603-615. doi: 10.1152/japplphysiol.00219.2024. Epub 2024 Jul 15. PMID 39008618
- [Background] Volpe D, Giantin MG, Maestri R, Frazzitta G. Comparing the effects of hydrotherapy and land-based therapy on balance in patients with Parkinson's disease: a randomized controlled pilot study. Clin Rehabil. 2014 Dec;28(12):1210-7. doi: 10.1177/0269215514536060. Epub 2014 Jun 3. PMID 24895382
- [Background] Hande D, Shinde S, Dhumale A, Kale HY. Effects of Aquatic-Based Resistance, Balance, and Proprioceptive Training on Ankle-Foot Malalignments in Postmenopausal Obese Women. Cureus. 2025 Jul 8;17(7):e87571. doi: 10.7759/cureus.87571. eCollection 2025 Jul. PMID 40786333
- [Background] Li Y, Zhuang R, Zhang J, Liu X. The effect of different exercise training modes on improving quality of life in patients with Parkinson's disease: a network analysis. Front Neurol. 2025 Jul 2;16:1601080. doi: 10.3389/fneur.2025.1601080. eCollection 2025. PMID 40672448
- [Background] Pezzini JV, Trevisan DD, Dominiak Soares VH, Gauer LE, Lima MMS. Sleep Quality in Parkinson Disease: Clinical Insights and PSQI Reliability Assessment. Sleep Sci. 2024 Oct 23;18(2):e147-e154. doi: 10.1055/s-0044-1791235. eCollection 2025 Jun. PMID 40672893
- [Background] Berardi A, Galeoto G, Valente D, Conte A, Fabbrini G, Tofani M. Validity and reliability of the 12-item Berg Balance Scale in an Italian population with Parkinson's disease: A cross sectional study. Arq Neuropsiquiatr. 2020 Jul;78(7):419-423. doi: 10.1590/0004-282X20200030. Epub 2020 Jun 8. PMID 32520233
- [Background] Petkus AJ, Foreman RP, Pilgrim M, Kim A, Hong E, Fisher BE, Van Horn JD, Wing D, Jakowec MW, Schiehser DM, Petzinger GM. Longitudinal associations between physical performance and cognition in individuals with Parkinson's disease. Clin Park Relat Disord. 2025 Jul 17;13:100370. doi: 10.1016/j.prdoa.2025.100370. eCollection 2025. PMID 40756809
- [Background] Yilmaz M, Atik-Altinok Y, Seyidoglu Yuksel D, Acarer A, Bozkurt D, Savas S, Sarac ZF, Akcicek F. Evaluation of sarcopenia and phase angle in elderly patients with Parkinson's Disease. Int J Neurosci. 2025 Apr;135(4):488-495. doi: 10.1080/00207454.2024.2310180. Epub 2024 Feb 1. PMID 38275120
- [Background] Villafane JH, Valdes K, Buraschi R, Martinelli M, Bissolotti L, Negrini S. Reliability of the Handgrip Strength Test in Elderly Subjects With Parkinson Disease. Hand (N Y). 2016 Mar;11(1):54-8. doi: 10.1177/1558944715614852. Epub 2016 Jan 14. PMID 27418890
- [Background] Cugusi L, Manca A, Bergamin M, Di Blasio A, Monticone M, Deriu F, Mercuro G. Aquatic exercise improves motor impairments in people with Parkinson's disease, with similar or greater benefits than land-based exercise: a systematic review. J Physiother. 2019 Apr;65(2):65-74. doi: 10.1016/j.jphys.2019.02.003. Epub 2019 Mar 21. PMID 30904467
- [Background] Yang Y, Wang G, Zhang S, Wang H, Zhou W, Ren F, Liang H, Wu D, Ji X, Hashimoto M, Wei J. Efficacy and evaluation of therapeutic exercises on adults with Parkinson's disease: a systematic review and network meta-analysis. BMC Geriatr. 2022 Oct 21;22(1):813. doi: 10.1186/s12877-022-03510-9. PMID 36271367
- [Background] Gamborg M, Hvid LG, Dalgas U, Langeskov-Christensen M. Parkinson's disease and intensive exercise therapy - An updated systematic review and meta-analysis. Acta Neurol Scand. 2022 May;145(5):504-528. doi: 10.1111/ane.13579. Epub 2022 Jan 8. PMID 34997759